CLINICAL TRIAL: NCT03956147
Title: Cultural Adaptation, Validation and Reability of the Munich Shoulder Questionnaire Into Turkish Patients With Shoulder Dysfunction
Brief Title: "Validation and Reability of the Munich Shoulder Questionnaire Into Turkish Patients"
Acronym: MSQ
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Deniz KOCAMAZ, principial investigator, Hasan Kalyoncu University
Other Study IDs: HEK12/224
Record Dates: First submitted 2019-04-16; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Shoulder Impingement; Shoulder Pain; Shoulder Injury
Keywords: Cultural adaptation; validation; responsibility; shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain; Shoulder Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Munich Shoulder Questionnaire — Validation and Reability study
  Other Names: Disability of arm, shoulder and hand; shoulder pain and disability index

SUMMARY:
The purpose of this study was to translate and culturally adapt the MSQ to Turkish language and test the validity and reliability of Turkish version of MSQ in shoulder dysfunction patients. And also, the ultimate goal was to facilitate international researches in shoulder problems as well as to serve the physicians for their clinical practice.

DETAILED DESCRIPTION:
Munich Shoulder Questionnaire (MSQ) is an innovative tool for self-assessment of shoulder function. It was especially designed for an effective follow-up of shoulder patients which were also allowing for a quantitative assessment of the Constant, Shoulder Pain and Disability Index (SPADI) and DASH score consisting of a 30-items questionnaire. It based on subjective and objective parameters of shoulder function.

Standart questionnaire enable to follow patients on a close and regular base with manageable effort for both the disability and the patients.an optimal instrument for outcome measurement of shoulder problems should meet the following requirments: a) the instrument should be a self-assmment patient reporting tool, b) the questions must be easily comprensible, c) filling in should be finished less than 30 minutes, d) the results should provide calculation of several well established scoring system. MSQ can be completed at home and typical functional abilities about evaluation are explained with pictures so these can make it easy. As a result, we choose to translate the MSQ into Turkish as it is less costly, practical and time consuming than developing a new tool. In addition, objective (normal joint movement and muscle strength) and subjective (pain, daily life activity, sport and leisure time activities) parameters in a single form to create the advantage in terms of ease of use and time. With these properties, MSQ may be preferred during follow-up of the results of conservative and / or surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* being between 18-65 years old,
* having unilateral or bilateral shoulder dysfunction,
* ability to read and complete the self-assessment questionnaires

Exclusion Criteria:

* have neurological, psychological and cardiovasculer diseases or injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: shoulder dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Objective and Subjective Items | 2 days
  The Munich Shoulder Questionnaire is a 30-items self-assessment questionnaire. Its raw score ranges from 0 to 314. For comparability, the raw numbers are divided by 314 giving a percentage ranging from 0 to 100 in which higher scores represent a better function of the shoulder.

SECONDARY OUTCOMES:
Objective Function | 2 days
  The objective function of the shoulder and consists of six items. The first five questions assess the range of motion: flexion, abduction, internal rotation, external rotation and range of the hand. Each question offer result from 0 to 10 points resulting in a total score ranging from a minimum of 0 to a maximum of 50 points ( 16 % of totals of MSQ) . The 6th targets at the power of the shoulder in 90° of abduction and 20° of quested to lift flexion. The patient is asked to fill a bag with items of daily living with a defined weıght such as a 500 gr water plastic bottle or bag. Then the patient is requested to lift the bag to the horizontal plane and hold 5 seconds. This is performed stepwise with increasing weights until the 12 kg. Each 500 gr is 2 point and maximum points is 24 for this question.(8%of the total MSQ).Altogether the objective part is a total score ranging from 0 to 74 points (%24 of the MSQ).
Subjective Function | 2 days
  subjective function and consists of 24 items. Six of the items deal with pain, nine cover work and activities of daily living, six cover sports and recreation activities and three ask for the social and emotional quality of life. This section accounts for a total score ranging from 0 to 240 points (%76 of the MSQ). It raw score ranges from 0 to 314. For comparability, the raw numbers are divided by 314 giving a percentage ranging from 0 to 100 in which higher scores represent a better function of shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ekici, Prof., Study Director — Hacettepe University
Locations (2):
- Turkey (Türkiye) (2):
  - Deniz Kocamaz, Gaziantep
  - Deni̇z Kocamaz, Gaziantep

IPD SHARING:
Plan to Share IPD: Yes
Validation and Reability of the Munich Shoulder Questionnaire Into Turkish Patients
Supporting Information: SAP
Time Frame: 3 months
Access Criteria: 18-65 years Having shoulder problem

REFERENCES:
- [Result] Yao M, Yang L, Cao ZY, Cheng SD, Tian SL, Sun YL, Wang J, Xu BP, Hu XC, Wang YJ, Zhang Y, Cui XJ. Chinese version of the Constant-Murley questionnaire for shoulder pain and disability: a reliability and validation study. Health Qual Life Outcomes. 2017 Sep 18;15(1):178. doi: 10.1186/s12955-017-0752-3. PMID 28923113
- [Result] Yuguero M, Huguet J, Griffin S, Sirvent E, Marcano F, Balaguer M, Torner P. Transcultural adaptation, validation and assessment of the psychometric properties of the spanish version of the Western Ontario Shoulder Instability Index questionnaire. Rev Esp Cir Ortop Traumatol. 2016 Nov-Dec;60(6):335-345. doi: 10.1016/j.recot.2016.07.003. Epub 2016 Aug 21. English, Spanish. PMID 27553522